CLINICAL TRIAL: NCT02568033
Title: Stereotactic Radiosurgery and Systemic Dose Chemotherapy for Locally Advanced Lung Cancer (Protocol Number GK001)
Brief Title: Stereotactic Radiosurgery and Systemic Dose Chemotherapy for Locally Advanced Lung Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-130
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Cisplatin; Docetaxel; Paclitaxel; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Chemotherapy:
  for Non-Squamous Cell: Pemetrexed 500 mg/m2 and cisplatin 75 mg/m2 on day 1 of 21 day cycle or Carboplatin AUC6 and Paclitaxel 75 mg/m2 on day 1 of 21 day cycle
  for Squamous Cell: Cisplatin 75 mg/m2 and docetaxel 75mg m2 day 1 of 21 day cycle or Carboplatin AUC6 and paclitaxel 200 mg/m2 day 1 of 21 day cycle
  Radiation- Stereotactic radiosurgery Peripheral Lung lesion: 60 Gy over 3 fractions Central Lung lesion: 50 Gy over 5 fractions Hilar and Mediastinal LNs 40-50Gy over 5 fractions
  Schedule is:
  2 cycles of chemotherapy, followed by SRS, followed by 2 additional cycles of chemotherapy.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: Docetaxel; Drug: Paclitaxel; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Drug: Pemetrexed
  Other Names: Alimta
Drug: Carboplatin
Drug: Cisplatin
Drug: Docetaxel
  Other Names: taxotere
Drug: Paclitaxel
  Other Names: taxol
Radiation: stereotactic radiosurgery
  Other Names: CK, cyberknife, cyber knife

SUMMARY:
This is a pilot study looking at using stereotactic radiosurgery and full dose chemotherapy to treat stage II and III lung cancer that is not amendable to surgical resection.

DETAILED DESCRIPTION:
Current standard of care for treatment of locally advanced (unresectable stage II and all of stage III) non-small cell lung cancer (NSCLC) is chemo-radiation which consists of 7 weeks of radiation and chemotherapy given at a reduced dose (as opposed to systemic dose when chemotherapy given by itself). While outcomes have improved over time they remain humbling, with current approaches associated with overall poor results both in terms of local (30% of patients have local failure) and distant control (40% of patients have distant failure) with a median overall survival of 17 months.

This study is evaluating treatment with full dose chemotherapy and stereotactic body radiotherapy (SBRT). SBRT uses high doses of radiation in a very precise and conformal manner, the number of treatments are much reduced versus conventional radiation (SBRT would be able to be completed in 2 weeks or less). The biologically effective dose of SBRT is much higher than that of conventional radiation; despite being a shorter number of treatments the effective radiation dose is higher. SBRT would be completed in 2 weeks and since radiation would be completed in a shorter time span, would allow patients to have higher (systemic) chemotherapy doses.

The purpose of this study is to explore SBRT in addition to systemic doses of chemotherapy in the treatment of locally advanced NSCLC.

ELIGIBILITY:
Inclusion criteria:

* Nonsmall cell lung cancer (NSCLC) (any histology)
* unresectable stage II
* Stage III
* Tumor less than 8 cm
* Karnofsky performance scale (KPS) of 50 or better
* Three or fewer mediastinal or hilar lymph nodes

Exclusion criteria

* Small cell lung cancer (SCLC)
* Stage I and stage IV patients
* Stage II patients eligible for surgical resection
* Concurrent severe disease that the treating physician feels will interfere with therapy this can include significant cardiovascular or pulmonary disease.
* KPS 40 or less (bed bound)
* Tumor size greater than 8 cm
* Inability to safely treat target lesions (at discretion of treating physician, this would most likely be secondary to not being able to place fiducial markers for tracking)
* Four or more medisatinal or hilar lymph nodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Disease free progression | 4-6 months
  Local control will be evaluated at end of treatment (4-6 months) and then at regular follow up intervals.
Toxicity (Treatment related side effects) | 4-5 months
  Treatment related side effects will be monitored

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center at Cooper, Camden, New Jersey, United States

REFERENCES:
- [Derived] Kubicek GJ, Khrizman P, Squillante C, Callahan K, Xu Q, Abouzgheib W, Boujaoude Z, Patel A, Hageboutros A. Stereotactic Body Radiotherapy and Systemic Dose Chemotherapy for Locally Advanced Lung Cancer: Single Arm Phase 2 Study. Am J Clin Oncol. 2022 Mar 1;45(3):129-133. doi: 10.1097/COC.0000000000000892. PMID 35195562